CLINICAL TRIAL: NCT04324567
Title: Inflammation After Laparoscopic Robot-assisted Surgery for Locally Advanced Rectal Cancer
Acronym: APR-IMM
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Ebbe Billmann Thorgersen, Principal Investigator, Oslo University Hospital
Other Study IDs: 2019/810
Record Dates: First submitted 2020-03-05; First posted 2020-03-27 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Locally Advanced Rectal Cancer; Abdominoperineal Resection
Keywords: Microdialysis; Inflammatory Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peritoneal fluid - daily samples as long as a pelvic drain is indicated. Regularly standard blood samples. Daily EDTA-plasma until post operative day 4, or longer if clinically indicated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- APR-open: Patients with locally advanced rectal cancer treated with neoadjuvant (chemo-) radiotherapy (CRT) and operated with abdominoperineal resection (APR) with laparotomy.
- APR-robot: Patients with locally advanced rectal cancer treated with neoadjuvant (chemo-) radiotherapy (CRT) and operated with abdominoperineal resection (APR) with laparoscopic robot assisted technique.

SUMMARY:
The intention of the study is to explore metabolic and inflammatory parameters in the pelvis and systemically after abdominoperineal resection (APR) for locally advanced rectal cancer (LARC) in patients that have received radiation therapy before surgery. In this study the inflammatory response after laparoscopic robot-assisted APR for LARC will be compared to results obtained in a recent cohort of patients operated with open APR for LARC, which will serve as the control population.

DETAILED DESCRIPTION:
Locally advanced rectal cancers (LARC) threaten the normal surgical margins and therefore needs neoadjuvant (chemo-) radiotherapy to down-stage the tumor before surgery. The Norwegian Radium Hospital Oslo University Hospital is a regional center for treatment of LARC in the south-eastern part of Norway and treat approximately 80-100 patients in this category annually. About 50 of these patients receive abdominoperineal resection (APR) as the main surgical treatment.

Laparoscopic surgery in LARC has been limited because of difficult dissection with straight instruments outside the normal anatomical planes in the confined space of the pelvis. However, recent papers report on better feasibility and good results in robot-assisted surgery for LARC. In respect to shorter postoperative length of stay for minimally invasive compared to open surgery, reduced inflammation may be the explanation, however, results are not conclusive. Most studies comparing open to minimally invasive surgery in colorectal cancer have had conventional laparoscopy as the minimally invasive group, including studies comparing inflammation after surgery. A study on inflammation after laparoscopic robot-assisted major surgery for bladder cancer has recently been published, but to our knowledge no comprehensive studies have been done with patients with rectal cancer resections. Additionally, there are claims that excessive and/or dysregulated inflammatory response after cancer surgery, worsen oncologic outcome. The need to characterize the inflammatory response after laparoscopic robot-assisted surgery of rectal cancer is thus highly relevant and needed.

The investigators want to analyse inflammatory parameters in plasma and peritoneal fluid in patients undergoing robot-assisted and open surgery for LARC.

Microdialysis is a technique which enables close to real-time monitoring of the tissues and organs of interest. The investigators want to utilize the microdialysis method to describe and monitor metabolic and inflammatory parameters in some patients after extensive robot-assisted oncological surgery for LARC.

The investigators hypothesize inflammatory response differ between patients undergoing open versus robot-assisted surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary rectal adenocarcinoma that have received radiation ≥25 Gy to the pelvis.
* operation with APR with laparoscopic robot assisted technique.
* have accepted and signed the consent form.

Exclusion Criteria:

* APR for other reasons

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer who receive radiotherapy >25 Gy prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Peak value of surgically induced C-reactive protein (CRP), expected to occur 1-3 days after surgery | December 2022
  CRP will be measured prior to surgery as well as on a daily basis the first 4 postoperative days. Peak values of CRP will be compared between patients undergoing open versus robot-assisted surgery.

SECONDARY OUTCOMES:
Overall survival at 1 year follow up after surgery | December 2024
  Differences between patients undergoing open versus robot-assisted surgery will be registered.
Progression-free survival at 1 year follow up after surgery | December 2024
  Differences between patients undergoing open versus robot-assisted surgery will be registered
Operating time in minutes | December 2023
  Differences between patients undergoing open versus robot-assisted surgery will be registered
Hospital length of stay in days after primary surgery | December 2023
  Differences between patients undergoing open versus robot-assisted surgery will be registered
Postoperative deep pelvic surgical site infection within 30 days after primary surgery | December 2023
  Differences between patients undergoing open versus robot-assisted surgery will be registered. Clinical diagnose (yes/no) supported by CT-scan
Superficial wound infection within 30 days after primary surgery | December 2023
  Differences between patients undergoing open versus robot-assisted surgery will be registered. Clinical diagnose (yes/no)
Dehiscence of the perineal wound at 3 months follow-up | December 2023
  Differences between patients undergoing open versus robot-assisted surgery will be registered. Clinical diagnose (yes/no)

OTHER OUTCOMES:
Monitoring inflammatory mediators in blood after neoadjuvant CRT and subsequent APR for LARC. | December 2023
  Blood be analysed using a multiplex cytokine assay (Bio-Plex Human Cytokine 27-Plex Panel, Bio-Rad Laboratories Inc., Hercules, CA). The following cytokines, chemokines and growth factors will be measured (all in pg/mL): Activated complement component 5 (C5a) Interleukin (IL) 1 beta (IL-1β), IL-1 receptor antagonist (IL-1Ra), IL-2, IL-4, IL-5, IL-6, IL-7, IL-8 (CXCL8), IL-9, IL-10, IL-12p70, IL-13, IL-15, IL-17, Eotaxin (CCL11), basic fibroblast growth factor (bFGF), granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon gamma (IFNG), interferon gamma inducible protein-10 (IP-10 or CXCL10), monocyte chemoattractant protein-1 (MCP-1 or CCL2), macrophage inflammatory protein-1-alpha (MIP-1α or CCL3), macrophage inflammatory protein-1-beta (MIP-1β or CCL4), platelet-derived growth factor-BB (PDGF-BB), regulated upon activation, normal T cell expressed and secreted (RANTES or CCL5), TNF-α and VEGF.
Monitoring inflammatory mediators in pelvic drain fluid after neoadjuvant CRT and subsequent APR for LARC. | December 2023
  Blood be analysed using a multiplex cytokine assay (Bio-Plex Human Cytokine 27-Plex Panel, Bio-Rad Laboratories Inc., Hercules, CA). The following cytokines, chemokines and growth factors will be measured (all in pg/mL): Activated complement component 5 (C5a) Interleukin (IL) 1 beta (IL-1β), IL-1 receptor antagonist (IL-1Ra), IL-2, IL-4, IL-5, IL-6, IL-7, IL-8 (CXCL8), IL-9, IL-10, IL-12p70, IL-13, IL-15, IL-17, Eotaxin (CCL11), basic fibroblast growth factor (bFGF), granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon gamma (IFNG), interferon gamma inducible protein-10 (IP-10 or CXCL10), monocyte chemoattractant protein-1 (MCP-1 or CCL2), macrophage inflammatory protein-1-alpha (MIP-1α or CCL3), macrophage inflammatory protein-1-beta (MIP-1β or CCL4), platelet-derived growth factor-BB (PDGF-BB), regulated upon activation, normal T cell expressed and secreted (RANTES or CCL5), TNF-α and VEGF.
Monitoring intermediate metabolites in the remnant muscular tissue of the pelvis floor in up to 10 patients with microdialysis catheters after neoadjuvant CRT and subsequent APR for LARC. | December 2023
  Lactate (mM), pyruvate (µM), lactate/pyruvate ratio, glycerol (µM) and glucose (mM) will be measured in microdialysis fluid from catheters inserted in the remnant muscular tissue of the pelvis floor after neoadjuvant CRT and subsequent APR for LARC to detect deep pelvic surgical site infection. The results will be compared to current standard monitoring. The measures will be done bedside on Iscus analyzer, M Dialysis AB, Stockholm, Sweden. The Iscus analyzer will calculate the lactate/pyruvate ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Ebbe B Thorgersen, MD PhD, Principal Investigator — Surgeon, The Department of Gastroenterological Surgery, The Norwegian Radium Hospital, Oslo University Hospital
Locations (1):
- The Norwegian Radium Hospital Oslo University Hospital, Oslo, Norway